CLINICAL TRIAL: NCT03051204
Title: OptiCal Study -Optimizing Fecal Calprotectin Monitoring: a Clinical Study Comparing CalproLab Against PhiCal and Evaluating Its Association With the Gut Microbiome
Acronym: OptiCal
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Genova Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB#16-001499
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Crohn Disease; Ulcerative Colitis; Irritable Bowel Syndrome; Celiac Disease; Healthy
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Irritable Bowel Syndrome; Celiac Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Aims:

To analyze stool specimens to test and validate the CalproLab assay against the predicate PhiCal in order to determine performance characteristics.

And to correlate Calpro levels to the gut microbiome composition.

DETAILED DESCRIPTION:
Fecal Calprotectin has become one of the most frequently used biomarkers in patients suffering from Inflammatory Bowel Diseases. Although its use for monitoring disease activity and therapeutic efficiency has previously been demonstrated, the test performance should further be optimized to improve clinical accuracy. The PhiCal™ test is a quantitative ELISA for measuring, in human stool, concentrations of fecal calprotectin, a neutrophilic protein that is a marker of mucosal inflammation. The PhiCal™ test can be used as an in vitro diagnostic to aid in the diagnosis of inflammatory bowel diseases (Crohn's disease and Ulcerative Colitis), and to differentiate IBD from irritable bowel syndrome. Recently, the CalproLab™ in vitro device has become available which provides a greater reporting range than PhiCal™. The OptiCal study aims to test and validate the CalproLab™ assay against the PhiCal™ assay and determine its performance characteristics.

Calprotectin is a valuable clinical marker for inflammation. Calprotectin belongs to a group of calcium- binding neutrophil-derived proteins. Calprotectin makes up 60% of the cytosolic proteins within the neutrophil. It is very resistant to bacterial degradation in the gut and is stable in stool for up to one week

at room temperature. Calprotectin is the noninvasive "test of choice" for quantifying the degree of GI inflammation and differentiating Irritable Bowel Syndrome (IBS) from Inflammatory Bowel Disease (IBD).

Inflammatory bowel disease (IBD) is considered to result from interplay between host and intestinal microbiota. Recently it was shown that the microbiota varied along a gradient of increasing intestinal inflammation (indicated by calprotectin levels), which was associated with reduced microbial richness, abundance of butyrate producers, and relative abundance of Gram-positive bacteria (especially Clostridium clusters IV and XIVa). A significant association between microbiota composition and inflammation was indicated by a set of bacterial groups predicting the calprotectin levels. So, intestinal microbiota may represent a potential biomarker for correlating the level of inflammation and therapeutic responses but this needs to be further validated.

* This study is a prospective case series during which patients with either Crohn's disease or ulcerative colitis, Celiac Disease, Irritable Bowel Syndrome and healthy controls (N=175) will be invited to participate.
* Participants will receive a home kit (with a plain white plastic cup for calprotectin sample collections) for stool sampling, which then will be returned and processed at Genova Diagnostics. All participants are required to complete a patient survey, which will be included in the collection kit.
* Participants will be recruited through the UCLA Division of Digestive Diseases.
* All patients will have confirmation of their diagnosis according to published clinical guidelines and standards of care using gold standard diagnostics (e.g. endoscopy)
* Stool specimens will be analyzed for fecal Calprotectin using both the CalproLab™ assay and the PhiCal™ assay. No blood draws or other testing will be performed.
* Patients will undergo a gut microbiome assessment utilizing the GI Effects™ 2200 Comprehensive Profile (Genova Diagnostics).

ELIGIBILITY:
Inclusion Criteria:

* Male and female IBD patients should have had CD or UC for at least a period of six months*
* Male and female patients should have had Celiac disease for at least three months.
* Subjects willing and able to sign informed consent
* Subjects willing and able to provide stool sample using a home kit
* IBS patients will meet Rome Foundation criteria and received standard of care evaluations to exclude other diagnoses
* Healthy controls will consist of patients who do not have any IBD or IBS diagnosis and meet exclusion criteria for health in nearby table

Exclusion Criteria:

* Unwilling or unable to adhere to the protocol
* Unwilling or unable to adhere to the informed consent
* Age <4y or >65y
* Any of the following conditions by medical history:

  * Individuals with intestinal cancer
  * Individual taking anti-inflammatory drugs
  * Individuals receiving chemotherapy
  * Individuals with a known intestinal infection
  * Individuals with known upper gastrointestinal disease such as esophagitis or gastritis that might influence the test's ability to detect intestinal inflammatory disease.
  * Individuals who are scheduled for endoscopy within 24 hours after providing the sample, or have undergone endoscopy during the 72 hours before providing the sample.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects 4-65y years of age with diagnosed Crohn's disease and ulcerative colitis.
  (75) IBD patients - Ulcerative Colitis (UC) or Crohn's Disease (CD) (50) IBS patients (25) Celiac Disease Patients (25) Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Calprotectin | up to 2 weeks from consent/enrollment
  Concentration of calprotectin in stool sample

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hommes, MD, Principal Investigator — UCLA IBD CENTER
Locations (1):
- UCLA Center for Inflammatory Bowel Diseases, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
All participants data will be de-identified by the research coordinator in standing with HIPAA regulations.